CLINICAL TRIAL: NCT05102110
Title: Feasibility Study to Investigate the Genomic and Epigenetic Changes in Rectal Mucus in Non-Colorectal Cancers of the Aero-Digestive Tract (ORI-EGI-03).
Brief Title: Feasibility Study to Investigate Rectal Mucus in Aero-Digestive Tract Cancer.
Acronym: ORI-EGI-03
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Origin Sciences (Industry)
Collaborators: Royal Devon and Exeter NHS Foundation Trust (Other)
Responsible Party: Sponsor
Other Study IDs: ORICOL-EGI-03
Record Dates: First submitted 2021-10-19; First posted 2021-11-01 (Actual); Last update posted 2024-08-05 (Actual); Status verified 2024-01

CONDITIONS: Non Small Cell Lung Cancer; Pancreatic Cancer; Bladder Cancer; Colorectal Cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Pancreatic Neoplasms; Urinary Bladder Neoplasms; Colorectal Neoplasms

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Rectal mucus collection with fragments of genetic material retrieved from rectal mucus.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Non-small cell lung cancer: A cohort of patients with known NSCLC who are assessed.
  Interventions: Diagnostic Test: Oricol Test
- Pancreatic cancer: A cohort of patients with known pancreatic adenocarcinoma who are assessed.
  Interventions: Diagnostic Test: Oricol Test
- Urothelial cancers: A cohort of patients with known uroepithelial cancers who are assessed.
  Interventions: Diagnostic Test: Oricol Test
- Colorectal cacncers: A cohort of patients with known colorectal cancers have been added to the study following methodology change in analysis techniques.

INTERVENTIONS:
Diagnostic Test: Oricol Test — Assessment of rectal mucus for material from aero-digestive cancers.
  Groups: Non-small cell lung cancer; Pancreatic cancer; Urothelial cancers

SUMMARY:
The aim of the study is to assess the feasibility of genomic and epigenetic analysis of rectal mucus to detect non-colorectal cancers of the aero- digestive tract using samples collected by the OriCol™ Sampling Device.

The primary objective of the study is to assess whether significant changes in DNA mutation and methylation associated with Non-colorectal cancers of the Aero- digestive Tract (NCRCADT) can be detected in rectal mucus as shed cells and cell-free DNA (cfDNA) pass through the gut and theoretically can be collected from rectal mucus.

Secondary objectives will assess the participant acceptability of the OriCol™ Sampling Device for Upper GI and Lung Pathology as well as contributing to a genomic library collating information about rectal mucus.

DETAILED DESCRIPTION:
The embryological development of the aero-digestive tract (ADT) is from a single primitive layer, the endoderm. Differentiation of this layer leads to epithelial and mucosal histopathological similarities through a continuous connected lumen extending from the upper third of the oesophagus to the anorectal junction and including the organs of the gastrointestinal tract (liver, pancreas, gallbladder) and the respiratory tract (trachea, bronchi and lung).

Cancers of the aero-digestive tract include; non-small cell lung (NSCLC), distal oesophageal, gastric, pancreatic, biliary, small bowel and colorectal cancer. The predominant type of cancer is an adenocarcinoma arising in the glandular cells lining the viscera. These cells have the capacity to secrete mucus and form the inner lining of the lumen All of these cancers directly or indirectly sheds cells into the gastrointestinal tract. The gastrointestinal epithelium regenerates every 5-7 days, the discarded cellular material migrates distally and is excreted as part of faeces. The majority of lung secretions are swallowed creating an interaction with the intestine which, to date, has primarily been studied from the microbiota perspective.

The Covid-19 pandemic has highlighted the strain on traditional diagnostic pathways, with a drop by 90% of the normal endoscopy workload in the first wave of the pandemic emphasising the need for practical investigations that can be used as a triage tool in primary care to discriminate individuals that do not require more invasive diagnostic tests. Rectal mucus sampling is potentially an appealing screening tool; quick, minimally invasive, cost effective, can be serially repeated for potential prognostic value, requires minimal equipment or training, and produces robust DNA material for extraction.

Recent research has demonstrated that stable, good quantity and quality cfDNA from colorectal cancer can be detected by rectal mucus sampling and clinical trials of the technique in symptomatic participants are underway looking at the use of rectal mucus for detection of colonic cancers (ClinicalTrials.gov, NCT identifier: NCT04659590). This unpublished, research has created a genomic profile of colorectal cancer in the rectal mucus using Next Generation Sequencing (NGS) detection of genetic mutations and alterations in methylation, which correlates with the documented genetic mutations associated with colorectal cancer tumour biopsies. Due to the embryological similarities KRAS and p53 are also found in association with other cancers of the GI tract. Discovered in 1983, methylation is a growing field in epigenetics, it is faster and more cost- effective than genetic mutation detection and promises increased sensitivity and specificity. The literature suggests a strong link between methylation changes and tumuorigenesis in cancers of the aero-digestive tract, which solely, or in conjunction with cf-DNA mutation detection, could play a significant role in early diagnosis.

This research aims to provide a novel insight into rectal mucus. The literature unanimously agrees that further research and standardisation of biomarkers and sampling is required. With novel genomic and epigenetic understanding of diagnostic and therapeutic targets a future of personalised oncological care is anticipated.

ELIGIBILITY:
Inclusion Criteria:

Aged 18 years or over Be able to give voluntary, written informed consent to participate in the study

Exclusion Criteria:

Participants with symptoms that would make proctoscopic examination inappropriate, including acute anal fissure, symptomatic thrombosed haemorrhoids or obstructing anorectal lesions as determined by rectal examination Participants with a previous history of cancer Participants who have received previously radiotherapy, chemotherapy or immunotherapy for a malignancy.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants with confirmed Non-small Cell Lung Cancer (NSCLC), Oesophageal, Gastric and Duodenal Cancer, Pancreatic Cancer, Biliary Tract Cancer (BTC) who have received a diagnosis but not commenced treatment at the time of participation.
  Control population will be participants with confirmed Urothelial Cancers who have received a diagnosis but not commenced treatment at the time of participation and participants with no known malignant pathology who have undergone a negative colonoscopy.
Sampling Method: Probability Sample
Enrollment: 450 (Estimated)
Dates: Start 2021-12-01 (Actual); Primary Completion 2025-06-30 (Estimated); Study Completion 2025-12-01 (Estimated)

PRIMARY OUTCOMES:
Correlation of SNP allele frequency in genes associated with known aero-digestive cancers in paired samples of tumour type and rectal mucus. | 1 year
  Genomic analysis

CONTACTS AND LOCATIONS:
Overall Officials: Mr F McDermott, FRCS, Study Director — Chief Investigator
Locations (1):
- Royal Devon & Exeter NHS Foundation Trust, Exeter, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided
Dependent upon initial sampling data.